CLINICAL TRIAL: NCT04780477
Title: Fiber-rich Foods to Treat Obesity and Prevent Colon Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Terry Hartman, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00000563; R01CA245063 (NIH)
Record Dates: First submitted 2021-03-02; First posted 2021-03-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Colon Cancer; Obesity
Keywords: Fiber-rich Foods; Legumes; Weight loss; Intestinal health; Cancer prevention
MeSH Terms: conditions — Colonic Neoplasms; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fiber Diet Featuring Legumes (HLD) (Experimental): Participants randomized to the high fiber diet featuring legumes (HLD) will add approximately 30 grams of dietary fiber per day from legume dishes, ensuring a total intake of approximately 50 grams of dietary fiber per day.
  Interventions: Dietary Supplement: High Fiber Diet Featuring Legumes (HLD)
- Healthy American Diet Control Arm (Active Comparator): Participants randomized to the healthy American diet control arm will receive pre-portioned meal replacement entrées with legumes replaced by lean chicken or meat.
  Interventions: Dietary Supplement: Healthy American Diet

INTERVENTIONS:
Dietary Supplement: High Fiber Diet Featuring Legumes (HLD) — The high fiber diet featuring legumes (HLD) provides pre-portioned entrées for two meals per day in months 1-3, and one meal per day in months 4-6. Participants continue on the diet in months 7-12 but assume responsibility for food preparation. The HLD will contain approximately 250 grams (g) of legumes per day (~1 ½ cups cooked legumes) in months 1-3 provided in two pre-portioned single serving entrées (i.e. ~125g in each serving). A study nutritionist provides in-person and written guidance for including side dishes that are nutritionally balanced with energy intake to lose 1-2 pounds of weight per week.
  Arms: High Fiber Diet Featuring Legumes (HLD)
Dietary Supplement: Healthy American Diet — The healthy American diet provides pre-portioned meal replacement entrées with legumes replaced by lean chicken or meat. Participants continue on the diet in months 7-12 but assume responsibility for food preparation. A study nutritionist provides in-person and written guidance for including side dishes that are nutritionally balanced with energy intake to lose 1-2 pounds of weight per week.
  Arms: Healthy American Diet Control Arm

SUMMARY:
This study tests whether a high-fiber diet based on legumes, such as dry beans, can lead to sustained reductions in obesity and colon cancer risk in persons at highest risk, namely overweight or obese, post-polypectomy patients.

DETAILED DESCRIPTION:
An important knowledge gap concerns the role of fiber in sustaining reduced energy intake to simultaneously manage weight and influence human colorectal cancer risk. Epidemiologic studies have shown an association between a high fiber diet featuring legumes (HLD) and reduced obesity and lower risk for adenoma recurrence or colorectal cancer. There are many plausible mechanisms to explain why high-fiber diets, and especially a HLD, may reduce colorectal cancer risk. First, fiber is fermented by the colonic microbiota to produce short chain fatty acids (SCFA). The SCFA, butyrate, has a remarkable array of colonic mucosal health promoting, anti-inflammatory, and anti-neoplastic properties. Secondly, microbiota break down plant cell walls releasing phytochemicals, which also have powerful anti-inflammatory and anti-carcinogenic effects. Thirdly, colonic transit is accelerated, reducing contact time with luminal carcinogens, such as heterocyclic amines formed from cooked red meat, and secondary bile acids, induced by a high fat diet and synthesized by the colonic microbiota.

Dr. Stephen O'Keefe's lab performed a human randomized controlled crossover feeding study (participants receive both diets) comparing high and low- fiber diets. The study measured mucosal biomarkers of cancer risk (proliferation - % epithelial cells staining positive for Ki67, inflammation - cluster of differentiation 3 (CD3)+ intraepithelial lymphocytes, cluster of differentiation 68 (CD68)+ lamina propria macrophages) made by fecal sampling and colonoscopy. Results suggested that within weeks these markers responded favorably to the high-fiber diet with proliferative rates and inflammatory biomarkers decreasing and microbiota composition adapting to increase butyrogenesis.

The researchers of this study have previously found that fiber may also reduce cancer risk indirectly by promoting weight loss, improving insulin sensitivity and decreasing inflammation. On average, individuals consume a similar weight of food daily; thus, replacing energy dense foods (higher kcal/g, e.g., high fat) with lower energy density foods (lower kcal/g), like legumes, should potentiate weight control. Viscous fiber intake is associated with longer gastric emptying times which over time might contribute to postponing the next eating occasion. Diet may also induce changes in gut microbiome composition leading to negative energy balance. Emerging human evidence links the gut microbiome with insulin resistance, inflammation, and obesity and with adenomatous polyps and colon cancer. In this current study, characterizing gut motility, microbiome, and metabolome composition profiles that may influence weight loss and have a role in the prevention or recurrence of adenomas and colorectal cancer, will provide novel and potentially therapeutic information.

The goal of the research is to conduct a clinical trial featuring study-provided pre-portioned entrées and strategic nutritional instruction to guide participants to integrate legumes into a healthy high-fiber diet pattern. Participants will be provided two entrées per day during months 1 through 3, and one entrée per day during months 4 through 6. Participants will continue their diets during months 7 through 12 but will be responsible for food preparation. The research will target a population at high risk for colorectal cancer, overweight and obese participants with a history of a colon polyp in the past 3 years, to test whether a high-legume, high-fiber diet will simultaneously increase weight loss and suppress intestinal biomarkers of cancer risk compared to a control diet (healthy American). In addition, it will explore potential mechanisms through which the high-legume intervention diet facilitates weight loss and intestinal health.

ELIGIBILITY:
Inclusion Criteria:

* free-living adults 40 to 75 years old
* BMI 25-40 kg/m^2
* able to provide documentation confirming a colonoscopy within 3 years that found ≥1 adenoma >0.5 cm or a sessile serrated polyp (any)
* English speaking
* ambulatory, able to pick up food, participate in clinical exams and laboratory tests
* able to provide informed consent

Exclusion Criteria:

* serious and/or unstable medical condition as deemed by study physician
* history of colorectal cancer, bowel resection, polyposis syndrome, or inflammatory bowel disease
* smoked regularly in the past year
* dietary restrictions substantially limiting compliance (e.g., must be willing to be randomized to either diet)
* planning on substantially changing usual exercise behavior in the next 6 months
* regular or recent use of prescription medication that may alter inflammation markers or gut function as deemed by study physician
* pregnant women, breast feeding women, or women planning pregnancy within the year of active study participation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline, Month 6 (end of intense intervention)
  Body weight is measured (in pounds) on a regularly calibrated digital scale while wearing light clothing without shoes.
Change in Ki-67+ Level | Baseline, Month 6 (end of intense intervention)
  Mucosal biopsies are obtained to measure the colonic mucosal proliferative biomarker Ki-67+.

SECONDARY OUTCOMES:
Change in Body Weight During Maintenance Period | Month 6, Month 12
  Body weight is measured (in pounds) on a regularly calibrated digital scale while wearing light clothing without shoes.
Change in Ki-67+ Level During Maintenance Period | Month 6, Month 12
  Mucosal biopsies are obtained to measure the colonic mucosal proliferative biomarker Ki-67+.
Change in Gut Transit Time | Baseline, Month 6 (end of intense intervention)
  Gut transit time is assessed using an indigestible single-use SmartPill capsule, a receiver, and display software. The SmartPill capsules were discontinued and no longer available after 2023 so participants beginning after January 19, 2024 will not complete this assessment.
Change in Fasting Plasma Insulin Level | Baseline, Month 6, Month 12
  Fasting plasma insulin, a biomarker of insulin resistance, is measured by blood test.
Change in Fasting Plasma Glucose Level | Baseline, Month 6, Month 12
  Fasting plasma glucose, a biomarker of insulin resistance, is measured by blood test.
Change in Serum C-reactive Protein | Baseline, Month 6, Month 12
  Serum C-reactive protein, an indicator of systemic inflammation, is measured by blood test.
Change in CD3+ Intraepithelial Lymphocytes Count | Baseline, Month 6, Month 12
  CD3+ intraepithelial lymphocytes, a colonic mucosal inflammatory biomarker of colon cancer risk, is measured by mucosal biopsy.
Change in CD68+ Lamina Propia Macrophages Count | Baseline, Month 6, Month 12
  CD68+ lamina propia macrophages, a colonic mucosal inflammatory biomarker of colon cancer risk, is measured by mucosal biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Hartman, PhD, MPH, RD, Principal Investigator — Emory University
Locations (1):
- Rollins School of Public Health, Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant phenotypic data will be made available for sharing but limited to health/biomedical purposes including age, obesity status, presence of colon polyps and history of diabetes. The data will be coded and only the coded data set, and not the master list, will be shared.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be made available for sharing beginning 9 months and ending 36 months following publication of findings for this study.
Access Criteria: Proposals to share individual participant data should be directed to tjhartm@emory.edu. To gain access, requestors will need to sign a data access agreement.
  To meet NIH data sharing requirements selected data will be deposited in appropriate research data repositories (e.g., NIH Common Fund Metabolomics Workbench). For genomic data, all data generated by this project will be made publicly available through adequate public genomic data warehouses as appropriate to the data type (NCBI Short Read Archives, Gene expression omnibus, etc.). Sequence data will be screened for the presence of sequences from human and these will be removed from public submissions unless directed otherwise by the NIH. Our algorithms will be made available through publications and as standalone programs when this is feasible. All new genomic and microbiome datasets will be deposited in public databases.

REFERENCES:
- [Derived] Hartman TJ, Christie J, Wilson A, Ziegler TR, Methe B, Flanders WD, Rolls BJ, Loye Eberhart B, Li JV, Huneault H, Cousineau B, Perez MR, O'Keefe SJD. Fibre-rich Foods to Treat Obesity and Prevent Colon Cancer trial study protocol: a randomised clinical trial of fibre-rich legumes targeting the gut microbiome, metabolome and gut transit time of overweight and obese patients with a history of noncancerous adenomatous polyps. BMJ Open. 2024 Feb 5;14(2):e081379. doi: 10.1136/bmjopen-2023-081379. PMID 38316601

DOCUMENTS (1):
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04780477/ICF_000.pdf